CLINICAL TRIAL: NCT07243691
Title: Study on the Therapeutic Effect of Different Infusion Times of Tislelizumab on Postoperative High-risk Hepatocellular Carcinoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sir Run Run Shaw Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SRRSH2025-0391
Record Dates: First submitted 2025-09-08; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — tislelizumab; Infusions, Intravenous

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cohort 1 (Experimental): Tislelizumab: 200mg, intravenous infusion, Q3W
  Interventions: Drug: Tislelizumab: 200mg, intravenous infusion, Q3W

INTERVENTIONS:
Drug: Tislelizumab: 200mg, intravenous infusion, Q3W — Postoperative adjuvant therapy (maximum of 8 cycles, each cycle lasting 21 days):
  - Tislelizumab: 200 mg, intravenous infusion, Q3W.
  Based on previous preclinical and clinical studies on circadian rhythms and adaptive immune responses, blood samples will be collected from patients at 05:00-07:00, 11:00-13:00, 17:00-19:00, and 23:00-01:00 (every 6 hours) to analyze the subset classification of peripheral blood lymphocytes. This will help map the immune circadian rhythm and determine the optimal injection time (which will then be used as the dosing time).

SUMMARY:
Study on the therapeutic effect of different infusion times on tislelizumab in high-risk postoperative hepatocellular carcinoma

ELIGIBILITY:
Inclusion Criteria:

1. (1) 18~75 years old (including boundary values).
2. (2) The first diagnosis confirmed by histology or cytology is HCC.
3. (3) Barcelona Clinical Liver Cancer (BCLC) stage A-B has undergone curative resection of the tumor, with no extrahepatic metastasis or adjacent organ invasion before surgery.
4. (4) Must meet at least one of the high-risk recurrence risk criteria (as follows): Characteristics of high-risk recurrent liver cancer after surgery: preoperative single lesion>5cm; MVI positive; Preoperative presence of sub lesions; Intraoperative margin<1cm.
5. (5) After one month of postoperative follow-up, there was no recurrence and no systemic treatment for HCC (systemic chemotherapy, immunotherapy, targeted therapy, or other treatments for HCC) was received.
6. (6) The Child Pugh score for liver function is 5-6 points, and the liver function is grade A.
7. (7) The physical fitness status score of the Eastern Cancer Collaboration Group (ECOG) is ≤ 1.
8. (8) Research on organ function levels that meet the requirements before the first use of medication; The functional indicators of important organs meet the following requirements: serum total bilirubin ≤ 51.3 μ mol/L or 3 mg/dL; Hemoglobin ≥ 90g/L, neutrophil count ≥ 1.5 × 10/L, platelet count ≥ 100 × 10/L; aspartate or alanine aminotransferase ≤ 5 times the upper limit of normal (ULN), alkaline phosphatase ≤ 2.5 ULN, serum albumin ≥ 30g/L; Serum creatinine<1.5 ULN; International normalized ratio (INR) ≤ 2 or prothrombin time (PT) exceeding the upper limit of the normal range ≤ 6 seconds; Serum creatinine ≤ 1.5 ULN, creatinine clearance rate ≥ 60 mL/min.
9. (9) Women who have the ability to conceive (i.e. physically capable of pregnancy) must agree to take effective contraceptive measures during the study period and within 120 days after the last dose of Trastuzumab treatment, and test negative for pregnancy within 7 days before the first dose of the study drug; Men who are capable of reproduction must agree to take effective contraceptive measures during the study period and within 120 days after the last administration of Trastuzumab.
10. (10) If the subject is infected with HBV or HCV The following conditions must be met: for inactive/asymptomatic HBV carriers, in the chronic phase; Active HBV (HBV deoxyribonucleic acid (DNA)<500 IU/mL (or 2500 copies/mL) during screening) should be treated according to treatment guidelines. Patients receiving antiviral therapy during screening should receive treatment>2 weeks prior to screening and continue treatment during the study period. For subjects infected with HCV: Confirmation of infection is based on detectable HCV ribonucleic acid RNA, and antiviral treatment must be completed before enrollment.
11. (11) The expected lifespan is ≥ 6 months.
12. (12) Voluntarily participate in this study and sign an informed consent form. If the subject does not have the ability to read the informed consent form (such as illiterate subjects), a witness must witness the informed process and sign the informed consent form.

Exclusion Criteria:

1. (1) The pathological diagnosis is non hepatocellular carcinoma.
2. (2) Within one month after surgery, there may be intrahepatic or extrahepatic recurrence.
3. (3) Previously received anti-tumor treatment plans such as chemotherapy, radiotherapy, radiofrequency ablation, interventional therapy, targeted therapy, and immunotherapy for liver cancer (excluding previous non tumor related surgeries and diagnostic biopsies).
4. (4) The viral load is limited to hepatitis B virus (HBV) DNA>2500 copies/ml, hepatitis C virus (HCV) RNA>1000, and no treatment has been received.
5. (5) Long term hormone users require long-term systemic hormone therapy (equivalent to>10 mg prednisone/day) or any other form of immunosuppressive therapy.
6. (6) Within the first 3 months of enrollment, there has been clinically significant bleeding or bleeding tendency, or ongoing thrombolytic or anticoagulant therapy.
7. (7) Patients with complete intestinal obstruction and those with incomplete intestinal obstruction in need of treatment (but those who relieve obstruction through fistula or stent placement can be included).
8. (8) Active severe clinical infections (>grade 2, NCI-CTCAE V5.0), including: active tuberculosis; Having a history of active tuberculosis infection for more than 1 year prior to enrollment; Has not received formal anti tuberculosis treatment or tuberculosis is still active.
9. (9) History of active immunodeficiency or autoimmune disease and/or possible recurrence of immunodeficiency or autoimmune disease in the past or long-term use of steroids.
10. (10) Uncontrolled diabetes (fasting blood glucose ≥ 10 mmol/L), severe lung disease (such as acute lung disease, pulmonary fibrosis affecting lung function, interstitial lung disease, but the recovered radiation pneumonia is excluded).
11. (11) Clinically significant cardiovascular diseases; Suffering from hypertension, antihypertensive drugs cannot effectively control (systolic blood pressure ≥ 140 mmHg or diastolic blood pressure ≥ 90 mmHg).
12. (12) Renal replacement therapy providers.
13. (13) Individuals who have allergic reactions to any component of the investigational drug.
14. (14) Within the past 5 years or currently suffering from other malignant tumors (excluding cured cervical carcinoma in situ, uterine carcinoma in situ, and non melanoma skin cancer).
15. (15) Pregnant or lactating female patients, and patients of childbearing age who refuse to receive contraceptive measures.
16. (16) Vulnerable groups, including individuals with mental illness, cognitive impairment, critically ill patients, etc.
17. (17) The researchers believe that patients who are not suitable to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-11-01 (Estimated); Study Completion 2027-12-15 (Estimated)

PRIMARY OUTCOMES:
2-year recurrence-free survival (RFS) rate | 2year

SECONDARY OUTCOMES:
recurrence-free survival (RFS) | From date of surgery until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months
  Duration from surgery to the first recorded HCC recurrence or all-cause death (whichever occurs first)
Time to recurrence (TTR) | From date of randomization until the date of first documented progression, assessed up to 36 months
  Defined as the time from enrollment to the first recorded disease recurrence assessed by the investigator,including the occurrence of local, regional, or metastatic HCC.
Overall survival (OS) | From date of surgery until the date of death from any cause, whichever came first, assessed up to 36 months
  Time from surgery to date of death, irrespective of cause.
1-year recurrence-free survival (RFS) rate | 1 year
1-year overall survival (OS) rate | 1year
2-year overall survival (OS) rate | 2year

OTHER OUTCOMES:
The incidence, severity, and correlation with the investigational product of adverse events (all adverse events, treatment emergent adverse events, serious adverse event) | 2year

CONTACTS AND LOCATIONS:
Locations (1):
- Sir Run Run Shaw Hospital, Zhejiang University School of Medicine (Qingchun Campus) 3 Qingchun Road East, Shangcheng District, Hangzhou, Zhejiang, China, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No